CLINICAL TRIAL: NCT06632717
Title: Efficacy and Safety of Hepatic Arterial Infusion Chemotherapy With Cisplatin and Fluorouracil in Combination With Lipiodol Embolization in Advanced Hepatocellular Carcinoma - a Prospective, Single-arm, Phase 2 Pilot Study
Brief Title: Hepatic Arterial Infusion Chemotherapy With Lipiodol Embolization in Advanced Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202311007MINA
Record Dates: First submitted 2024-07-10; First posted 2024-10-09 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatic Arterial Infusional Chemotherapy; Lipiodol Embolization; Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Cisplatin; Fluorouracil; Ethiodized Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAIC-Cisplatin+5-fluorouracil in combination with lipiodol embolization (Experimental): hepatic arterial infusional cisplatin and 5-fluorouracil will be given followed by lipiodol embolization
  Interventions: Drug: Cisplatin; Drug: 5-fluorouracil; Procedure: Lipiodol embolization

INTERVENTIONS:
Drug: Cisplatin — Chemotherapy regimen
  • Cisplatin 60mg/m2 on day 2; 5-fluorouracil (5-FU) 500mg/m2 on day 1 - day 3 via the HAIC port, every 3 weeks until progression or intolerable toxicity
Drug: 5-fluorouracil — Chemotherapy regimen
  • Cisplatin 60mg/m2 on day 2; 5-fluorouracil (5-FU) 500mg/m2 on day 1 - day 3 via the HAIC port, every 3 weeks until progression or intolerable toxicity
  Other Names: 5-FU
Procedure: Lipiodol embolization — Lipiodol embolization protocol
  * Lipiodol embolization will be performed on day 3 after completion of 5-FU infusion, up to 4 cycles. Fixed dose lipiodol of 10mL will be given on day 3 followed by 30mL normal saline flush.
  * The administration of lipiodol is mandatory on cycle 1. The administration of lipiodol on cycle 2 to cycle 4 will depend on the discretion of the treating physician and the presence of adverse effects from lipiodol embolization.
  Other Names: ethiodized oil

SUMMARY:
Hepatic artery infusion chemotherapy (HAIC) is a locoregional therapy commonly used in hepatocellular carcinoma (HCC), with high response rates and minimal impairment of liver function reported. Transarterial chemoembolization (TACE) and transarterial embolization (TAE) are also commonly used in HCC, with high response rates reported yet carry risks of impairing liver function after repeated embolization with a definitive embolic agent. On the other hand, lipiodol used in TACE/TAE has transient and plastic embolization effects on the tumor in contrast to the long-lasting embolization effect of the definitive embolic agent. This study investigates whether combining HAIC with lipiodol embolization will increase efficacy with good liver function preservation.

DETAILED DESCRIPTION:
Hepatic artery infusion chemotherapy (HAIC) is an effective locoregional therapy commonly utilized in hepatocellular carcinoma (HCC). The rationale for the anti-tumor efficacy of HAIC is to deliver high local concentrations of chemotherapeutic agents to the liver tumor. Previous studies on HAIC alone or in combination with other systemic therapies have demonstrated excellent intrahepatic tumor contr rates and survival benefits. The investigators have previously conducted a pilot study of HAIC in National Taiwan University Hospital (NTUH) using cisplatin and 5-fluorouracil and demonstrated a high response rate of 26% in advanced HCC patients. In addition to the observed efficacy, HAIC does not impair liver function significantly over repeated administration and can be safely given to patients with poor or limited liver reserve.

Transarterial chemoembolization (TACE) and transarterial embolization (TAE) are the most recognized standard treatment in intermediate-stage HCC and are also commonly utilized in advanced-stage HCC. TACE procedure is based on administering a cytotoxic drug mixed with lipiodol followed by definitive embolization of the tumor-feeding arteries by an embolic agent. However, repeated embolization can impair liver function and jeopardize the chance of patients receiving further salvage treatment. Lipiodol used in TACE/TAE has transient and plastic embolization effects on the tumor in contrast to the long-lasting embolization effect of the embolic agent, such as Gelfoam. Performing embolization with lipiodol alone without an embolic agent may limit detrimental effects on the normal liver and help preserve liver function in patients with HCC.

The investigators hypothesize that combining HAIC and transient embolization using lipiodol may have enhanced efficacy compared to HAIC alone. In addition, the unwanted liver function impairment caused by repeated embolization is alleviated by the characteristic transient embolization effect of lipiodol. Thus, The investigators propose this prospective, single-arm, phase 2 pilot study comprising HAIC with cisplatin and 5-fluorouracil in combination with lipiodol embolization to investigate its efficacy and safety in patients with advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF).
2. Histologically or clinically (typical HCC imaging findings by multi-phase CT or MRI) diagnosed HCC.
3. Barcelona Clinic Liver Cancer (BCLC) Stage C disease (liver confined disease or liver predominant disease, as determined by the investigator) or BCLC Stage B disease who failed standard treatment (i.e., TACE in intermediate stage HCC or systemic therapy in advanced HCC) or refused standard treatment or intolerable to standard treatment.
4. Archival tissue available (< 2 years) or agree to have biopsy tissue at baseline
5. Age > 20 years at the time of study entry.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. Child-Pugh class A or B7
8. ≥1 measurable lesion per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 in the liver
9. Body weight >30 kg
10. Adequate normal organ and marrow function as defined below:

(1) Hemoglobin ≥9.0 g/dL (2) Absolute neutrophil count (ANC) ≥1.0 x 109/L (≥ 1,000 per mm3) (3) Platelet count ≥75 x 109/L (≥75,000 per mm3) (4) Serum bilirubin ≤2 x institutional upper limit of normal (ULN). (5) AST (SGOT)/ALT (SGPT) ≤3x institutional upper limit of normal unless active liver malignancies are present, in which case it must be ≤5x ULN (6) Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance: 11. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.

12. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

13. Must have a life expectancy of at least 12 weeks

Exclusion Criteria:

1. Fibrolamellar carcinoma or mixed hepatocellular cholangiocarcinoma
2. The result of lung perfusion scan of the HAIC port > 30%
3. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
4. Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies) ≤14 days prior to the first dose of the study drug. If sufficient wash-out time has not occurred due to the schedule or PK properties of an agent, a longer wash-out period will be required, as agreed by the principal investigator.
5. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.
6. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
7. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of study treatment.
8. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection (except HBV infection or HCV infection), symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
9. History of another primary malignancy except for conditions listed in the protocol.
10. History of leptomeningeal carcinomatosis
11. Brain metastases or spinal cord compression. Patients with suspected brain metastases at screening should have an MRI (preferred) or CT each preferably with IV contrast of the brain prior to study entry
12. History of active primary immunodeficiency
13. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice)
14. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of the trial treatment.
15. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (RECIST 1.1) | From date of randomization until the date of first documented confirmed response rate by RECIST 1.1, assessed up to 60 months
  To assess the objective response rate (RECIST 1.1) of HAIC-PF + lipiodol embolization.

SECONDARY OUTCOMES:
Objective response rate (mRECIST) | From date of randomization until the date of first documented confirmed response rate by mRECIST, assessed up to 60 months
  To assess the objective response rate (modified RECIST) of HAIC-PF + lipiodol embolization
Liver specific objective response rate (RECIST 1.1 & modified RECIST) | From date of randomization until the date of first documented liver specific confirmed response rate by RECIST 1.1 & mRECIST, assessed up to 60 months
  To assess the liver specific objective response rate (RECIST 1.1 & modified RECIST) of HAIC-PF + lipiodol embolization.
Progression-free survival (RECIST 1.1 and modified RECIST) | From date of randomization until the date of first documented progression (RECIST 1.1 or mRECIST) or date of death from any cause, whichever came first, assessed up to 60months
  To assess the progression-free survival (RECIST 1.1 or modified RECIST) of HAIC-PF + lipiodol embolization
Overall survival | From date of randomization until the date of first documented date of death from any cause, whichever came first, assessed up to 60 months
  To assess the overall survival of HAIC-PF + lipiodol embolization
Incidence of treatment-emergent adverse events [safety and tolerability] | From date of randomization until 3 months after the end-of-trial, assessed up to 60months
  To assess the incidence of treatment-emergent adverse events of HAIC-PF + lipiodol embolization by reporting number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Tsung-Hao Liu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan